CLINICAL TRIAL: NCT00474630
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study Comparing the Safety and Efficacy of Naltrexone 32 mg Sustained Release (SR)/Bupropion 360 mg Sustained Release (SR) and Placebo in Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Safety and Efficacy Study Comparing Naltrexone SR/Bupropion SR and Placebo in Obese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NB-304; COR-Diabetes (Other: Orexigen Therapeutics, Inc.)
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Overweight; Diabetes Mellitus, Type 2
Keywords: Obesity; Overweight; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NB32 (Experimental): Naltrexone SR 32 mg/bupropion SR 360 mg/ day with ancillary therapy
  Interventions: Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/ day; Behavioral: Ancillary therapy
- Placebo (Placebo Comparator): Placebo with ancillary therapy
  Interventions: Drug: Placebo; Behavioral: Ancillary therapy

INTERVENTIONS:
Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/ day
  Other Names: NB32
  Arms: NB32
Drug: Placebo
  Arms: Placebo
Behavioral: Ancillary therapy — Ancillary therapy consisting of diet instruction, advice on behavior modification, and exercise counseling

SUMMARY:
The purpose of this study is determine whether the combination of naltrexone SR and bupropion SR is safe and effective in treating obesity in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Optimal care of patients with diabetes mellitus includes vigorous and persistent efforts to achieve physiologic control of blood glucose as well as other often associated conditions including hypertension, dyslipidemia and excess weight. Pharmacologic interventions for the treatment of obesity in type 2 diabetes have shown significant reductions in HbA1c. Two Phase II clinical trials demonstrated that a combination of bupropion SR and naltrexone is associated with greater weight loss than bupropion SR alone, naltrexone alone, or placebo in subjects with uncomplicated obesity. The current study investigated the safety and efficacy of the combination of naltrexone SR and bupropion SR compared to placebo in obese subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18 to 70 years of age (inclusive)
* Body mass index (BMI) ≥27 and ≤45 kg/m²
* Diagnosed with type 2 diabetes mellitus and on no injectable antidiabetes medication or inhaled insulin for more than 3 months prior to randomization
* Took stable doses of oral single or combination hypoglycemic medications (biguanides, thiazolidinediones, meglitinides, α-glucosidase inhibitors, sulfonylureas, DPP4 inhibitors) for at least 3 months prior to randomization or did not take medications for the treatment of type 2 diabetes mellitus
* Normotensive (systolic ≤145 mm Hg and diastolic ≤95 mm Hg). Antihypertensive medications were allowed with the exception of alpha-adrenergic blockers, and clonidine. Antihypertensive treatment was stable for at least 4 weeks prior to randomization.
* Medications for the treatment of dyslipidemia were allowed with the exception of cholestyramine and cholestypol as long as the medical regimen had been stable for at least 4 weeks prior to randomization.
* Free of opioid medication for 7 days prior to randomization
* HbA1c between 7% and 10%, fasting blood glucose <270 mg/dL, and fasting triglycerides <400 mg/dL
* No clinically significant abnormality of serum albumin, blood urea nitrogen (BUN), bilirubin, calcium, and phosphorus
* Creatinine levels were ≤1.4 mg/dL for female subjects and ≤1.5 mg/dL for male subjects
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels were within 2.5 × upper limit of laboratory normal range (ULN)
* No clinically significant abnormality of hematocrit, white blood cell (WBC) count, WBC differential, or platelets
* No clinically significant abnormality on urinalysis
* TSH within normal limits or normal T3, if TSH is below normal limits
* Female subjects of childbearing potential had a negative serum pregnancy test
* Negative urine drug screen
* An IDS-SR score <2 on individual items 5 (sadness), 6 (irritability), 7 (anxiety/tension), and 18 (suicidality) and an IDS-SR total score <30
* Female subjects of childbearing potential were non-lactating and agreed to continue to use effective contraception throughout the study and 30 days after discontinuation of study drug
* Able to comply with all required study procedures and schedule
* Able to speak and read English
* Provided written informed consent

Exclusion Criteria:

* Type I diabetes mellitus
* "Brittle-diabetes" or any hospitalization or emergency room visit due to poor diabetic control within 6 months prior to screening, history of diabetes-related dehydration leading to hospitalization, or history or evidence of ketoacidosis
* Obesity of known endocrine origin other than diabetes mellitus (e.g., untreated hypothyroidism, Cushing's syndrome, established polycystic ovary syndrome)
* Diabetes mellitus secondary to pancreatitis or pancreatectomy
* Serious medical condition including but not limited to renal or hepatic insufficiency and Class III or IV congestive heart failure; history of myocardial infarction, angina pectoris, claudication, or acute limb ischemia within 6 months prior to screening; lifetime history of stroke
* History of malignancy with exception of non-melanoma skin cancer or surgically cured cervical cancer within 5 years prior to screening
* Loss or gain of more than 5.0 kg within the 3 months prior to screening
* Severe microvascular or macrovascular complications of diabetes, including but not limited to proliferative retinopathy, active limb ulcerations, amputation of metatarsals or above
* Serious psychiatric illness, including lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, and anorexia nervosa; current serious personality disorder (e.g., borderline or antisocial); current severe major depressive disorder; recent (6 months prior to screening) suicide attempt or current active suicidal ideation; or recent hospitalization due to psychiatric illness
* Response to the bipolar disorder questions that indicated the presence of bipolar disorder
* Required medications for the treatment of a psychiatric disorder (with the exception of short term insomnia) within 6 months prior to screening
* History of drug or alcohol abuse or dependence within 1 year prior to screening
* Baseline ECG with a QTc interval (Bazett's formula) >450 msec (men) and >470 msec (women) or the presence of any clinically significant cardiac abnormalities, including but not limited to patterns consistent with recent myocardial ischemia, electrolyte abnormalities, or atrial or ventricular dysrhythmia or significant conduction abnormalities
* Received the following excluded concomitant medications: any psychotropic agents (including antipsychotic, antidepressant, anxiolytic, mood stabilizer, anticonvulsant agents, and agents for the treatment of attention deficit disorder) with the exception of low-dose benzodiazepine or hypnotic agents for the treatment of insomnia (up to 2 mg lorazepam/day or equivalent dose of a benzodiazepine or hypnotic agent); any anorectic or weight loss agents; any over-the-counter dietary supplements or herbs with psychoactive, appetite, or weight effects; alpha-adrenergic blockers; dopamine agonists; clonidine; coumadin; theophylline; cimetidine; oral corticosteroids; cholestyramine, cholestypol, Depo Provera®; smoking cessation agents; use of opioid or opioid-like medications, including analgesics and antitussives
* History of surgical or device intervention for obesity (e.g., gastric banding)
* History of seizures of any etiology, or of predisposition to seizures (e.g., history of cerebrovascular accident, head trauma with ≥5 minutes loss of consciousness, concussion symptoms lasting ≥15 minutes, brain surgery, skull fracture, subdural hematoma, or febrile seizures)
* Treatment with bupropion or naltrexone within 12 months prior to screening
* History of hypersensitivity or intolerance to bupropion or naltrexone
* Changes in smoking status or in tobacco or nicotine use within 3 months prior to screening or planned during study participation
* Participated in a weight loss management program within one month prior to randomization
* Females who were pregnant or breast-feeding or planned to become pregnant during the study period or within 30 days of discontinuing study drug
* Planned surgical procedure that could impact the conduct of the study
* Received any investigational drug or used an experimental device or procedure within the previous 30 days
* Participated in any previous clinical trial conducted by Orexigen
* Had any condition that in the opinion of the investigator made the subject unsuitable for inclusion into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - SelfCenter, PC, Fairhope, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - HealthStar Research, Hot Springs, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - Northern California Research, Carmichael, California
  - Sierra Medical Research, Fresno, California
  - Advance Clinical Research Institute, Orange, California
  - Affiliated Research Institute, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Apex Research Institue, Santa Ana, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - LCFP Inc., Fort Myers, Florida
  - Miami Research Associates, Miami, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - CSRA Partners in Health, Inc, Augusta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Deaconess Clinic, Evansville, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - L-Marc, Louisville, Kentucky
  - Trover Center for Clinical Studies, Madisonville, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Health Trends Research, LLC, Baltimore, Maryland
  - FutureCare Studies, Springfield, Massachusetts
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Center for Nutrition and Metabolic Diseases, Univ. of Nevada, Reno, Nevada
  - Endocrinology & Diabetes Consultants, Dover, New Hampshire
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Diabetes care and Information Center, Flushing, New York
  - Central New York Clinical Research, Manlius, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Central Ohio Nutrition Center, Inc., Columbus, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Your Diabetes Endocrine and Nutrition Group, Mentor, Ohio
  - Mountain View Clinical Research, Greer, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - The Cooper Institute, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Diabetes & Glandular Disease Research Associates, Inc., San Antonio, Texas
  - Summit Research Network, Inc., Seattle, Washington
  - Northside Internal Medicine, Spokane, Washington

REFERENCES:
- [Result] Hollander P, Gupta AK, Plodkowski R, Greenway F, Bays H, Burns C, Klassen P, Fujioka K; COR-Diabetes Study Group. Effects of naltrexone sustained-release/bupropion sustained-release combination therapy on body weight and glycemic parameters in overweight and obese patients with type 2 diabetes. Diabetes Care. 2013 Dec;36(12):4022-9. doi: 10.2337/dc13-0234. Epub 2013 Oct 21. PMID 24144653

RESULTS

PARTICIPANT FLOW:
Groups:
- NB32: Naltrexone SR 32 mg/Bupropion SR 360 mg/day
- Placebo: Placebo
Period: Overall Study
Arm/Group | NB32 | Placebo
Started | 335 | 170
Completed | 175 | 100
Not Completed | 160 | 70
Not completed — Adverse Event | 98 | 26
Not completed — Lost to Follow-up | 22 | 15
Not completed — Withdrawal by Subject | 21 | 15
Not completed — Protocol Violation | 3 | 4
Not completed — Lack of Efficacy | 5 | 6
Not completed — Drug noncompliance, other | 11 | 4

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | NB32 | Placebo | Total
Number analyzed (Participants) | 335 | 170 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.02 (9.05) | 53.46 (9.83) | 53.83 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 90 | 285
  Male | 140 | 80 | 220
Race/Ethnicity, Customized [Number; unit: participants]
  White | 261 | 140 | 401
  Black or African American | 63 | 18 | 81
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 2 | 2 | 4
  Other | 1 | 5 | 6
Weight [Mean (Standard Deviation); unit: kg] | 104.22 (18.93) | 105.08 (16.99) | 104.51 (18.28)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.40 (4.75) | 36.40 (4.50) | 36.40 (4.66)

OUTCOME MEASURES:

1. Primary Outcome: Co-primary: Body Weight- Mean Percent Change
Time Frame: Baseline, 56 weeks
Population: Modified ITT (Full Analysis Set): Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of body weight | -5.03 (0.34) | -1.75 (0.43)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.28, 95% CI [-4.34 to -2.22]

2. Secondary Outcome: Change in HbA1c Levels
Time Frame: Baseline, 56 weeks
Population: Modified ITT: Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent
Groups:
- NB32: Naltrexone SR 32 mg/bupropion SR 360 mg/ day
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 222 | 137
percent | -0.63 (0.07) | -0.14 (0.09)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.71 to -0.27]

3. Primary Outcome: Co-primary: Body Weight- Proportion of Subjects With ≥5% Decrease
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 44.53 [38.54 to 50.51] | 18.87 [12.79 to 24.95]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.44, 95% CI 2-sided [2.15 to 5.50]

4. Secondary Outcome: Change in Fasting Triglycerides Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 222 | 135
percent change | -11.20 [-15.59 to -6.58] | -0.80 [-6.95 to 5.76]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Net) = -10.4

5. Secondary Outcome: Change in Fasting HDL Cholesterol Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 222 | 135
mg/dL | 3.03 (0.49) | -0.29 (0.61)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.32, 95% CI 2-sided [1.80 to 4.84]

6. Secondary Outcome: Change in Fasting Blood Glucose Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 264 | 158
mg/dL | -11.87 (2.70) | -4.02 (3.39)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.065, ANCOVA; Mean Difference (Net) = -7.85, 95% CI 2-sided [-16.21 to 0.50]

7. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 208 | 124
cm | -4.97 (0.47) | -2.89 (0.61)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -2.08, 95% CI 2-sided [-3.57 to -0.59]

8. Secondary Outcome: Body Weight- Proportion of Subjects With ≥10% Decrease
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 18.49 [13.82 to 23.16] | 5.66 [2.07 to 9.25]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 3.75, 95% CI 2-sided [1.79 to 7.88]

9. Secondary Outcome: HbA1c- Proportion of Subjects With HbA1c <7% at Endpoint
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 222 | 137
percentage of participants | 44.14 [37.61 to 50.68] | 26.28 [18.91 to 33.65]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 2.46, 95% CI 2-sided [1.50 to 4.04]

10. Secondary Outcome: Percent of Subjects Requiring Rescue Medications for Diabetes
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 22.26 [19.05 to 29.91] | 35.22 [29.81 to 45.36]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.35 to 0.86]

11. Secondary Outcome: Percent of Subjects With Dose Reduction in Oral Antidiabetes Medications
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 1.89 [0.28 to 3.87] | 1.26 [0.00 to 3.19]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.27 to 7.57]

12. Secondary Outcome: Percent of Subjects With Dose Increase in Oral Antidiabetes Medications
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 3.02 [1.06 to 5.58] | 1.26 [0.00 to 3.19]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.55 to 12.67]

13. Secondary Outcome: Change in HOMA-IR Levels, Using Log-transformed Data
Description: HOMA-IR= Homeostasis Model Assessment-Insulin Resistance
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 199 | 112
percent change | -20.56 [-27.77 to -12.62] | -14.67 [-24.69 to -3.31]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -5.89

14. Secondary Outcome: Change in Fasting Insulin Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 201 | 113
percent change | -13.48 [-19.70 to -6.78] | -10.35 [-18.75 to -1.09]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -3.13

15. Secondary Outcome: HbA1c- Proportion of Subjects With HbA1c <6.5% at Endpoint
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 222 | 137
percentage of participants | 20.72 [15.39 to 26.05] | 10.22 [5.15 to 15.29]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.36 to 5.14]

16. Secondary Outcome: Change in IWQOL-Lite Total Scores
Description: IWQOL-Lite= Impact of Weight on Quality of Life-Lite Questionnaire Total score is based on a scale from 0 to 100, with 0 representing the poorest and 100 the best quality of life and where a score of 71-79 indicates moderate impairment
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 241 | 153
units on a scale | 9.27 (0.70) | 7.90 (0.86)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 1.37, 95% CI 2-sided [-0.77 to 3.51]

17. Secondary Outcome: Change in High-sensitivity C Reactive Protein (Hs-CRP) Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 202 | 119
percent change | -20.91 [-29.29 to -11.54] | -13.29 [-24.94 to 0.17]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -7.62

18. Secondary Outcome: Percent of Subjects Discontinuing Due to Poor Glycemic Control
Description: Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed. Odds ratio not calculated as there were no subjects in the NB32 group that discontinued due to poor glycemic control.
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
percentage of participants | 0 [NA to NA] — There were no subjects in the NB32 group that discontinued due to poor glycemic control. | 1.89 [0.00 to 4.00]

19. Secondary Outcome: Change in Question 19 From 21-Item COE (Control of Eating) Questionnaire
Description: Question 19: Generally, how difficult has it been to control your eating? Scoring: 0=not at all difficult; 100=extremely difficult
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 225 | 146
units on a scale | -11.89 (1.39) | -6.91 (1.69)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -4.98, 95% CI 2-sided [-9.22 to -0.74]

20. Secondary Outcome: Change in Fasting LDL Cholesterol Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 220 | 134
mg/dL | -1.44 (1.94) | -0.01 (2.44)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -1.43, 95% CI 2-sided [-7.48 to 4.62]

21. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
mm Hg | 0.03 (0.70) | -1.12 (0.88)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 1.16, 95% CI 2-sided [-1.02 to 3.33]

22. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
mm Hg | -1.06 (0.47) | -1.47 (0.59)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.41, 95% CI 2-sided [-1.04 to 1.86]

23. Secondary Outcome: Change in IDS-SR Total Scores
Description: IDS-SR= Inventory of Depressive Symptoms-Subject Rated IDS-SR total score is based on 30 items. The total score can range from 0-84, with 0 being no depressive symptoms and 84 being very severe depressive symptoms. A total score ≤ 13 indicates no depression.
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 265 | 159
units on a scale | 0.01 (0.33) | -1.60 (0.42)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 1.62, 95% CI 2-sided [0.59 to 2.65]

24. Secondary Outcome: Change in Food Craving Inventory Sweets Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The sweets subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 241 | 155
units on a scale | -1.97 (0.28) | -2.40 (0.34)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.43, 95% CI 2-sided [-0.42 to 1.27]

25. Secondary Outcome: Change in Food Craving Inventory Carbohydrates Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The carbohydrates subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 241 | 155
units on a scale | -1.48 (0.26) | -1.52 (0.32)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.04, 96% CI 2-sided [-0.76 to 0.85]

ADVERSE EVENTS:
Time Frame: Baseline, 56 weeks
Description: The safety analysis set includes all randomized subjects who took study drug and were assessed by investigator after their first dose, whether or not they discontinue the study. Treatment-emergent adverse events were defined as events that started or worsened in the double-blind treatment phase after the first dose and before 7 days post last dose.
Groups:
- NB32: Naltrexone SR 32 mg/Bupropion SR 360 mg daily
Arm/Group | NB32 | Placebo
Serious Adverse Events (participants affected / at risk) | 13/333 | 8/169
Other Adverse Events (participants affected / at risk) | 275/333 | 109/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=333) | Placebo (N=169)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=333) | Placebo (N=169)
Abdominal pain upper (Gastrointestinal disorders) | 17 (18) | 3 (4)
Constipation (Gastrointestinal disorders) | 59 (69) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 52 (60) | 16 (21)
Dry mouth (Gastrointestinal disorders) | 21 (22) | 5 (5)
Nausea (Gastrointestinal disorders) | 141 (196) | 12 (13)
Vomiting (Gastrointestinal disorders) | 61 (80) | 6 (7)
Oedema peripheral (General disorders) | 2 (3) | 10 (15)
Influenza (Infections and infestations) | 9 (9) | 9 (9)
Nasopharyngitis (Infections and infestations) | 28 (32) | 23 (25)
Sinusitis (Infections and infestations) | 16 (19) | 14 (19)
Upper respiratory tract infection (Infections and infestations) | 26 (30) | 16 (22)
Diabetes mellitus (Metabolism and nutrition disorders) | 15 (16) | 15 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 25 (65) | 12 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 12 (13)
Dizziness (Nervous system disorders) | 39 (52) | 9 (11)
Headache (Nervous system disorders) | 46 (53) | 15 (18)
Tremor (Nervous system disorders) | 22 (26) | 4 (4)
Anxiety (Psychiatric disorders) | 18 (20) | 2 (2)
Insomnia (Psychiatric disorders) | 37 (42) | 9 (10)
Hypertension (Vascular disorders) | 33 (33) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 18 months after conclusion of the study at all study centers, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 60 days to review and comment on the proposed publication. The review period may be extended by an additional 30 days upon request. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.